CLINICAL TRIAL: NCT03689348
Title: Acute and Chronic (28 Days) Effects of Avena Sativa Extract on Physiological and Psychological Responses to Stress, and Mood and Cognitive Function
Brief Title: Acute and Chronic Effects of Avena Sativa on Cognition and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Anklam Extrakt (Industry)
Responsible Party: Principal Investigator, Emma Wightman, Principal investigator, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 57BV1
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Cognitive Change; Stress, Psychological; Mood
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Maltodextrin powder is the placebo ingredient and this is encased in the same pale green capsules as the active ingredient. Participants, if in the placebo group, will consume x3 capsules of placebo per day for 28 days.
  Interventions: Dietary Supplement: Placebo
- 300mg Avena sativa (Experimental): If in the 300mg of Avena sativa group, participants will consume x2 placebo capsules (described above) and x1 300mg capsule of Avena sativa per day for 28 days.
  Interventions: Dietary Supplement: Avena sativa
- 600mg Avena sativa (Experimental): If in the 600mg of Avena sativa group, participants will consume x1 placebo capsule (described above) and x2 300mg capsule of Avena sativa per day for 28 days.
  Interventions: Dietary Supplement: Avena sativa
- 900mg Avena sativa (Experimental): If in the 300mg of Avena sativa group, participants will consume x3 300mg capsule of Avena sativa per day for 28 days.
  Interventions: Dietary Supplement: Avena sativa

INTERVENTIONS:
Dietary Supplement: Avena sativa — A supplement derived from wild green oat
  Other Names: Wild green oat
  Arms: 300mg Avena sativa; 600mg Avena sativa; 900mg Avena sativa
Dietary Supplement: Placebo — Maltodextrin
  Arms: Placebo

SUMMARY:
The flavanoid and terpene phytochemicals present in wild green oat interact with multiple mechanisms relevant to brain function; including those which would modulate cognition and stress. The current study aims to test this in a group of N=128 males and females between the ages of 35-65yrs before and after 28 days supplementation of placebo, 300-, 600- and 900mg of a wild green oat extract.

DETAILED DESCRIPTION:
The flavanoid and terpene phytochemicals present in wild green oat interact with multiple mechanisms relevant to brain function; including those which would modulate cognition and stress. The current study aims to test this in a group of N=128 males and females between the ages of 35-65yrs before and after 28 days supplementation of placebo, 300-, 600- and 900mg of a wild green oat extract. The study is randomized (within x3 age categories also; 35-45, 46-55, 56-65yrs), placebo controlled and counterballanced across parallel groups. Participants will first attend a training/screening session followed by x2 lab-based testing sessions, 28 days apart. In the lab-based sessions participants will complete baseline cognitive assessments; including whilst undergoing a stressful observed methodology (the observed multi-tasking stressor or 'OMS'). Here galvanic skin response and heart rate will be measured and before and after the OMS participants will provide a saliva sample which will be analysed for cortisol and alpha-amylase levels. This procedure will be repeated 120- and 240- minutes post-dose. Between the lab-based sessions participants will complete mood scales via a mobile phone application 'cognimapp'.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-assess themselves as being in good health
* Aged 35 to 65 years at the time of giving consent
* In employment and/or higher education or full time child-care

Exclusion Criteria:

Participants are not eligible to take part if they:

* Have any pre-existing medical condition/illness which will impact taking part in the study NOTE: the explicit exceptions to this are controlled (medicated) arthritis, asthma, hay fever, high cholesterol and reflux-related conditions. There may be other, unforeseen, exceptions and these will be considered on a case-by-case basis; i.e. participants may be allowed to progess to screening if they have a condition/illness which would not interact with the active treatments or impede performance.
* Are currently taking prescription medications NOTE: the explicit exceptions to this are contraceptive and hormone replacement treatments for female participants where symptoms are stable and treatment will not change during the course of the study, those medications used in the treatment of arthritis, high cholesterol and reflux-related conditions; and those taken 'as needed' in the treatment of asthma and hay fever. As above, there may be other instances of medication use which, where no interaction with the active treatments is likely, and which would not be expected to impede the participant's ability to perform the study assessments, participants may be able to progress to screening.
* Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
* Have a Body Mass Index (BMI) outside of the range 18.5-35 kg/m2
* If still menstruating/fertile, are pregnant, seeking to become pregnant or lactating. If undergoing menopause, are not stable on medication (no adverse symptoms) for at least the last 3 months
* Have learning and/or behavioural difficulties such as dyslexia or ADHD
* Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
* Smoker
* excessive caffeine intake (>500 mg per day)
* Have relevant food intolerances/ sensitivities
* Have taken antibiotics within the past 4 weeks
* Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Are unable to complete all of the study assessments
* Are currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks
* Has been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months
* Suffers from frequent migraines that require medication (more than or equal to 1 per month)
* Sleep disorders or are taking sleep aid medication
* Any known active infections
* Does not have a bank account (required for payment)
* Does not have access to the Internet (inc via smart phone)
* Are non-compliant with regards treatment consumption

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Changes in mood; as assessed by the 'Profile Of Mood States' (POMS) | Pre-dose and post-dose on day 1 and day 29
  Mood will be assessed with the profile of mood states questionnaire questionnaire and this will be completed at the start and end of the testing day on day 1 and day 29. To assess if the investigational product (IP) has changed mood a change score will be calculated (end of day minus start of day) and this will be compared between the x4 treatment groups.
Changes in mood; as assessed by the 'General Anxiety Disorder- 7' (GAD-7) questionnaire | Day 1, 8, 15, 22 and 29
  Mood will be assessed with the general anxiety disorder-7 questionnaire on day 1 and then again on day 8, 15, 22 and 29 of the study intervention period. Change from baseline scores will be calculated and, at each subsequent time point, scores will be compared across the x4 treatment groups to ascertain if the IP has changed mood.
Changes in mood; as assessed by the 'General Health Questionnaire' (GHQ) | Pre-dose and post-dose on day 1 and day 29
  Mood will be assessed with the general health questionnaire and this will be completed at the start and end of the testing day on day 1 and day 29. To assess if the investigational product (IP) has changed mood a change score will be calculated (end of day minus start of day) and this will be compared between the x4 treatment groups.
Changes in cognitive function | Pre-dose and 120 minutes and 240 minutes post-dose on day 1 and day 29
  Cognitive function will be assessed via several individual cognitive tasks (stroop, rapid visual information processing and corsi blocks) and will together provide indicators of accuracy and speed. This data will be collected at baseline, 120- and 240-minutes post-dose on day 1 and day 29. Change from baseline scores will be calculated and compared across the x4 treatment groups to ascertain if the IP has changed cognitive function.
Changes in subjective stress; as assessed by the 'perceived stress scale' (PSS) | Pre-dose and 120 minutes and 240 minutes post-dose on day 1 and day 29
  Subjective stress will be measured via the perceived stress scale before and after each completion of the observed multitasking stressor (OMS) on day 1 and on day 29. The change in the stress response between pre- and post-OMS will be compared across the x4 treatment groups to ascertain if the IP has changed subjective perceptions of stress.
Changes in subjective stress; as assessed by the 'state, trait anxiety inventory' (STAI) | Pre-dose and 120 minutes and 240 minutes post-dose on day 1 and day 29
  Subjective stress will be measured via the state, trait anxiety inventory before and after each completion of the observed multitasking stressor (OMS) on day 1 and on day 29. The change in the stress response between pre- and post-OMS will be compared across the x4 treatment groups to ascertain if the IP has changed subjective perceptions of stress.
Changes in objective stress; as assessed by salivary cortisol levels | Pre-dose and 120 minutes and 240 minutes post-dose on day 1 and day 29
  Saliva samples will be taken from participants before and after each completion of the observed multitasking stressor (OMS) and the change in salivary cortisol levels between pre- and post-OMS will be compared across the x4 treatment groups to ascertain if the IP has changed the objective stress response
Changes in objective stress; as assessed by salivary alpha-amylase levels | Pre-dose and 120 minutes and 240 minutes post-dose on day 1 and day 29
  Saliva samples will be taken from participants before and after each completion of the observed multitasking stressor (OMS) and the change in salivary alpha amylase levels between pre- and post-OMS will be compared across the x4 treatment groups to ascertain if the IP has changed the objective stress response
Changes in objective stress; as assessed by galvanic skin response (GSR) | Pre-dose and 120 minutes and 240 minutes post-dose on day 1 and day 29
  Galvanic skin response (GSR) will be recorded throughout the observed multitasking stressor (OMS) and the change in GSR across the OMS will be compared across the x4 treatment groups to ascertain if the IP has changed the objective stress response
Changes in objective stress; as assessed by heart rate (HR) | Pre-dose and 120 minutes and 240 minutes post-dose on day 1 and day 29
  Heart rate (HR) will be recorded throughout the observed multitasking stressor (OMS) and the change in HR across the OMS will be compared across the x4 treatment groups to ascertain if the IP has changed the objective stress response.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Wightman, Dr, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The IPD will be shared with the study sponsor (Anklam Extrakt) and the named investigators.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT03689348/Prot_SAP_001.pdf